CLINICAL TRIAL: NCT03876470
Title: Micro-elimination of Hepatitis C in a Rural Appalachian Community: The Implementation and Expansion of an Innovative Collaborative Care Model of Telehealth and Knowledge Sharing Focusing on People Who Inject Drugs
Brief Title: Conquering Hepatitis C Via Micro-Elimination in Southwest Virginia
Acronym: CHIME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Rebecca Dillingham, MD/MPH, Director of the Center for Global Health, University of Virginia
Other Study IDs: 21167
Record Dates: First submitted 2019-02-25; First posted 2019-03-15 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Telehealth; Injection Drug Use
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants will receive HCV treatment as determined by their provider. HCV treatment is not assigned by the study.
  Interventions: Other: Hepatitis C treatment as chosen by provider

INTERVENTIONS:
Other: Hepatitis C treatment as chosen by provider — Participants' providers will determine the type of HCV treatment as appropriate.

SUMMARY:
The objective of this protocol is to conduct a comprehensive quantitative and qualitative assessment of the impact of our innovative collaborative telehealth HCV care model on patient treatment experiences and quality of life.

DETAILED DESCRIPTION:
The investigators will evaluate the proportion of patients at each step of the HCV care cascade before and after implementation of the collaborative care model. Additionally, participants will complete questionnaires at three time points: at the initiation of hepatitis C treatment, at treatment completion, and at the assessment of sustained virologic response. Questionnaires will assess quality of life, mental health, chronic liver disease outcomes, and substance use. A subset of participants will also complete semi-structured interviews at each of the three time points. Then, a smaller subset of participants will be selected for a detailed ethnographic case study focusing on treatment experiences, quality of life, forms of social support, and illness experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Detectable HCV viral load
* Attended a clinic appointment at one of our participating sites

Exclusion Criteria:

* Cognitive disability such that informed consent cannot be obtained
* Prisoners
* Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 subjects will be enrolled. Of these, 20 will be enrolled in the qualitative interviews and 4 will be enrolled in the ethnographic case studies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Cohort-level Hepatitis C Treatment Progress | 12 months
  Change in the proportion of patients at each step of the HCV care continuum (linkage to care, treatment initiation, treatment completion and sustained virologic suppression) before and after program implemenation

SECONDARY OUTCOMES:
Patient Reported Quality-of-Life | 12 months
  Change in SF-12 scores from treatment initiation to treatment completion and sustained virologic response
Depression | 12 months
  Change in Patient Health Questionnaire-2 (PHQ-2) scores from treatment initiation to treatment completion and sustained virologic response. Scale range: 0 to 6 with a higher score indicative of greater depressive symptoms.
Health-Related Quality-of-Life | 12 months
  Change in Chronic Liver Disease Questionnaire: Hepatitis C version (CLDQ-HCV) scores from treatment initiation to treatment completion and sustained virologic response. Scores range from 1 to 7 with higher scores indicative of better quality of life. CLDQ-HCV includes a total score and 4 sub-scales (activity/energy, emotional, worry, and systemic), each scored from 1 to 7.
Semi-Structured Qualitative Interview about Impact of HCV Treatment | 12 months
  Qualitative assessment of participants' experience with HCV treatment, including its impact on substance use behaviors, activities of daily living, social interactions, and mental and physical health

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Dillingham, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No